CLINICAL TRIAL: NCT03343158
Title: Orphans and Vulnerable Children Risk Screening Tool Research Study (Zimbabwe)
Status: Terminated | Type: Observational
Why Stopped: Significantly more resources would have been necessary to complete the study.
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: JSI Research & Training Institute, Inc. (Other); Biomedical Research and Training Institute, Zimbabwe (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); World Education, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EG0174
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Orphans, Children, Adolescents; Vulnerable Children, Adolescents; Community-based

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators propose to assess the sensitivity, specificity, positive and negative predictive value of an HIV Risk Screening Tool in identifying the risk of being HIV-infected among Orphans and Vulnerable Children (OVC) aged 2-18 years in a community setting.

DETAILED DESCRIPTION:
In the first phase of the study, investigators will identify an optimal set of screening questions with acceptable sensitivity and false positive rate, based on the draft 11-question pilot tool. Using the identified questions, investigators will develop a composite screening tool and determine criteria that should be used for identifying children for testing with minimally acceptable sensitivity and false positive rates. In the second phase of the study, investigators will select optimal questions to create a composite screening tool and validate it in a similar study population. Investigators anticipate the accuracy of the tool will be much improved compared to the individual questions. Investigators will also assess the usability of the HIV Risk Screening Tool as measured by the time taken to administer the tool, and perceptions of its ease and simplicity.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents ages 2 up to 18 years living in a household and enrolled in WEI/Zimbabwe and/or partners program;
* Children/adolescents ages 2 up to 18 years with HIV status unknown, or who tested negative three or more months ago;
* Children/adolescents ages 2 up to 18 years who are healthy or ill (unless they are ill enough to require immediate hospitalization).

Exclusion Criteria:

* Children/adolescents aged 2 up to 18 years tested HIV positive
* Children/adolescents ages 2 up to 18 years who require immediate hospitalization;
* Children/adolescents ages 2 up to 18 years who refuse/are refused participation.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: OVC aged 2-18 years, living in households which are registered on a database developed by World Education Institute, a Non-Government Organization which provides services for orphans and vulnerable children in the community
Sampling Method: Probability Sample
Enrollment: 2260 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Phase 1: Validity of various questions in predicting the probability of HIV among OVC (Screening tool) | Four weeks
  Sensitivity and specificity of eleven questions in predicting HIV among OVC
Phase 2: Validation of combined questions in predicting HIV among OVC (Validating Screen tool) | Six weeks
  Validation of combined questions assessed from Phase 1 in predicting HIV among OVC

SECONDARY OUTCOMES:
Usability of screening tool | Two weeks
  CHWs who participate in the screening will be invited to participate in a short survey, offered in either Shona or English (depending on participant choice), on the ease, simplicity, and usability of the screening tool, as well as perceptions of the process

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Mahomva, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Godfrey Woelk, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- EGPAF Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No